CLINICAL TRIAL: NCT04473144
Title: The Effect of Ulistin on Acute Renal Injury in Patients Undergoing OPCAB (Off Pump Coronary Artery Bypass): a Propensity Score Matched Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, Assistant professor, Ajou University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MED-MDB_20-257
Record Dates: First submitted 2020-07-08; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — urinastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Anesthesia induction and maintenance and postoperative recovery management were performed according to the standard anesthesia protocol for off pump coronary artery bypass surgery.
- Ulistin (Sham Comparator): In the Ulistine administration group, 300,000 KIU was mixed with 100 mL physiological saline and administered over 15 minutes after induction of anesthesia.
  Anesthesia induction and maintenance and postoperative recovery management were performed according to the standard anesthesia protocol for off pump coronary artery bypass surgery.
  Interventions: Drug: Ulinastatin

INTERVENTIONS:
Drug: Ulinastatin — In the Ulistine administration group, 300,000 KIU was mixed with 100 mL physiological saline and administered over 15 minutes after induction of anesthesia.
  Arms: Ulistin

SUMMARY:
Acute kidney injury (AKI) is a frequent complication after cardiac surgery. AKI has been reported as 7-40% depending on the type of surgery, and is known to increase to about 50% when there are risk factors. Cardiac surgery-associated AKI (CSA-AKI) requires cardiac replacement therapy in 1-5% of patients and increases mortality to 1,4%, but the treatment is still unknown. Therefore prevention of occurrence is very important.

Known factors related to the development of CSA-AKI include hemodynamic, inflammatory, metabolic, and nephrotoxic factors, and since there is a close connection between hypotension due to deterioration of cardiac function, preventive measures to prevent hypotension in juicing It is only possible.

To date, strategies to protect kidneys with drugs are very limited. Urinary trypsin inhibitor, ulistine, has anti-inflammatory and antioxidant effects, so it has been reported to protect against renal ischemia/reperfusion injury. Various studies have been attempted to prevent CSA-AKI, but most of them are inflammatory reactions during surgery. It was performed only for surgery with extracorporeal circulation that causes severely.

Therefore, this study would like to verify the effectiveness of ulistine's medicine in the prevention of CSA-AKI in patients undergoing coronary artery bypass surgery without extracorporeal circulation.

ELIGIBILITY:
Inclusion Criteria:

* From January 2015 to June 2020, a retrospective study will be conducted on patients undergoing extracorporeal circulatory coronary artery bypass surgery at Ajou University Hospital.

Exclusion Criteria:

* Patients who were undergoing renal replacement therapy prior to surgery due to end-stage renal failure are excluded from the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of acute kidney injury | 7 days after operation
  Cr ≥ 0.3 mg/dl within 48 hours after surgery, 1.5 times higher preoperative value within 7 days, urine volume <0.5 ml/kg for 6 hours after surgery

IPD SHARING:
Plan to Share IPD: No